CLINICAL TRIAL: NCT01947595
Title: Prediabetes Lifestyle Intervention Study
Brief Title: Individualized Lifestyle Intervention in Subjects With Prediabetes
Acronym: PLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Diabetes-Center, Leibniz-Institut in Düsseldorf (Other); Endocrinology and Metabolic Diseases, Charité Berlin (Unknown); German Institute of Human Nutrition (Other); University Hospital Carl Gustav Carus (Other); LMU München, medical clinic IV (Unknown); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, andreas fritsche, Prof. Dr. med. Andreas Fritsche, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DZD-2012
Record Dates: First submitted 2013-06-25; First posted 2013-09-20 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes mellitus type 2; impaired glucose tolerance; lifestyle intervention; body fat distribution; prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

ARMS (4):
- high risk non-responder, intensified lifestyle intervention (Active Comparator): high risk non-responder:
  * A) reduced Insulin secretion (disposition index: (IGI * ISI-Matsuda)< 760)
  * B) insulin resistance (ISI-Matsuda < 9,2)
  * C) elevated liver fat ( MRT > 5,56%)
  * A+B or A+C or B+C or A+B+C
  Interventions: Behavioral: intensified lifestyle intervention
- hight risk non responder, normal lifestyle intervention (Active Comparator): high risk non-responder:
  * A) reduced Insulin secretion (disposition index: (IGI * ISI-Matsuda)< 760)
  * B) insulin resistance (ISI-Matsuda < 9,2)
  * C) elevated liver fat ( MRT > 5,56%)
  * A+B or A+C or B+C or A+B+C
  Interventions: Behavioral: normal lifestyle intervention
- Responder, normal lifestyle intervention (Active Comparator): Responder:
  * A) reduced Insulin secretion (disposition index: (IGI * ISI-Matsuda)< 760)
  * B) insulin resistance (ISI-Matsuda < 9,2)
  * C) elevated liver fat ( MRT > 5,56%)
  * No A, only B or C
  Interventions: Behavioral: normal lifestyle intervention
- Responder, single lifestyle advice (control group) (Active Comparator): Responder:
  * A) reduced Insulin secretion (disposition index: (IGI * ISI-Matsuda)< 760)
  * B) insulin resistance (ISI-Matsuda < 9,2)
  * C) elevated liver fat ( MRT > 5,56%)
  * No A, only B or C
  Interventions: Behavioral: Single lifestyle advice

INTERVENTIONS:
Behavioral: intensified lifestyle intervention — * physical activity 6 hours per week, 50% guided activity
    * recorded by an accelerometer (Aipermotion 440)
  * 16 sessions per year with a lifestyle advisor
    * nutritional advice (target weight: 5% less, if BMI > 25kg/m², less than 30% fat per caloric intake, less than 10% fatty acids per caloric intake, more than 15 g fibre per 1000 kcl)
  Arms: high risk non-responder, intensified lifestyle intervention
Behavioral: normal lifestyle intervention — * physical activity 3 hours per week
    * recorded by an accelerometer (Aipermotion 440)
  * 8 sessions per year with a lifestyle advisor
    * nutritional advice (target weight: 5% less, if BMI > 25kg/m², less than 30% fat per caloric intake, less than 10% fatty acids per caloric intake, more than 15 g fibre per 1000 kcl)
  Arms: Responder, normal lifestyle intervention; hight risk non responder, normal lifestyle intervention
Behavioral: Single lifestyle advice — - Single Health care advice and lifestyle advice (30 minutes) at the beginning
  * recommend the individual target weight (5% less, if BMI 25> kg/m²)
  Arms: Responder, single lifestyle advice (control group)

SUMMARY:
The purpose of this prospective randomized multicenter intervention study is to determine whether in the prevention of Diabetes an intensified lifestyle intervention is superior to a conventional lifestyle intervention in high risk non-Responder subjects. Further, the intensive phenotyping to determine subgroups with an increased risk for diabetes enables an individualized prevention and therapy of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The study start with an intensive phenotyping at baseline (initial examination) to determine subjects with prediabetes. These high risk non-Responder are randomized in two arms (intensified vs normal lifestyle intervention)with equal number of subjects (n=250). The results are compared with each other at the end of the study.

The low risk Responder are randomized in two arms (normal vs. once lifestyle intervention = control group) with equal number of subjects (n=250).

After the screening at baseline the 12 month lifestyle intervention starts for lifestyle intervention groups. The different therapy groups are formed as described before. The subjects with intensified lifestyle intervention get 16 consultations, the subjects with normal lifestyle intervention get 8 consultations, the subjects of the control group get one consultation to learn more about a healthier lifestyle. During the whole study there is a continuous supervision from physician and nutritional advisers and the subjects have to document a nutrition and an exercise protocol as well as subjective measurements. At baseline, after 24 weeks and at follow up 1, 2 and 3 years later there is an elaborate metabolic characterization of all subjects (also the Responder groups) a 75 g venous oral glucose tolerance test (OGTT) as well as an analysis of the distribution of body fat confirmed by MR-Imaging and proton magnetic resonance spectroscopy by 3 T whole body imager.

ELIGIBILITY:
Inclusion Criteria:

* impaired fasting glucose (IFG)

  * fasting blood glucose 99-126 mg/dl

and/or

* impaired glucose tolerance (IGT)

  * 75 g OGTT 120 minutes: 139-200 mg/dl

Exclusion Criteria:

* current pregnancy or breastfeeding
* BMI > 45 kg/m²
* Diabetes mellitus Typ 1 or 2
* serious disease e.g symptomatic coronary heart disease
* serious symptomatic malignant disease (weight loss > 10% within the last 6 month)
* severe liver or kidney disease ( an increase in transaminases > 3 times than the upper limit of the standardized range, GFR < 50 ml/min/1,73m²)
* systemic infection (CRP > 1 mg/dl)
* severe mental illness
* drug abuse
* treatment with steroids
* potentially incompliant subjects
* exclusion criteria for magnetic resonance tomography

  * any kind of metal in or on the body:

    * cardiac pacemakers
    * prosthetic heart valves
    * metal prosthesis
    * magnetic implanted metallic parts
    * contraceptive coil
    * metal fragments/ grenade shrapnel
    * fixed braces
    * acupuncture needles
    * insulin pump
    * intraport etc.
    * Field strength > 3 Tesla further tattoos, permanent make-up
  * persons with limited thermosensory or heightened sensitivity to heating
  * persons where cardiovascular disease cannot be ruled out by examination
  * persons with heightened sensitivity to loud noise or diseases of the ear
  * used closed whole body scanner: claustrophobia

Additional for spirometry

* acute coronary syndrome
* higher cardiac arrhythmia
* decompensated heart failure
* acute carditis
* pulmonary embolism
* acute deep leg vein thrombosis ( phlebothrombosis)
* hyperthyroidism (TSH)
* hypokalemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2012-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
postprandial glycaemia (2h plasma glucose level of the 75 g oral glucose tolerance test (OGTT)) | one year

SECONDARY OUTCOMES:
insulin sensitivity confirmed by 75 g oral glucose tolerance test (OGTT) | one year
  insulin resistance is calculated as follows:
  * Insulinogenic index (IGI) = (I30 - I0) / (G30 - G0)
  * ISIest= 10000/²√ ((G0 x I0) x ((G0+G30+G60+G90+G120)/5) x ((I0+I30+I60+I90+I120)/5))
insulin secretion confirmed by 75 g oral glucose tolerance test (OGTT) | one year
  insulin resistance is calculated as follows:
  * Insulinogenic index (IGI) = (I30 - I0) / (G30 - G0)
  * ISIest= 10000/²√ ((G0 x I0) x ((G0+G30+G60+G90+G120)/5) x ((I0+I30+I60+I90+I120)/5))
distribution of body fat confirmed by MR-Imaging and proton magnetic resonance spectroscopy by 3 T whole body imager | one year

OTHER OUTCOMES:
metabolic and genetic characterization to determine the risk of type 2 diabetes confirmed by case history, clinical examination, venous blood sampling, DNA isolation, standardised questionnaires, bio-electric impedance analysis (BIA)and ergospirometry | one year
metabolic and genetic characterization to determine the non-response to lifestyle intervention confirmed by case history, clinical examination, venous blood sampling, DNA isolation, standardised questionnaires,BIA, ergospirometry | one year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fritsche, Prof. Dr. med, Principal Investigator — University Hospital Tuebingen; Norbert Stefan, Prof.Dr.med., Principal Investigator — University Hospital Tübingen
Locations (7):
- Germany (7):
  - Deutsches Institut für Ernährungsforschung / Charité Berlin, Berlin
  - University Hospital Dresden, Dresden
  - Deutsches Diabetes Zentrum, Düsseldorf
  - Technische Universität München (TU Munich), Munich
  - Helmholtz Zentrum München, Munich
  - Ludwig-Maximilians-University, Munich
  - University Hospital Tübingen, Tübingen

REFERENCES:
- [Derived] Wagner R, Eckstein SS, Fritsche L, Prystupa K, Horber S, Haring HU, Birkenfeld AL, Peter A, Fritsche A, Heni M. Postprandial Dynamics of Proglucagon Cleavage Products and Their Relation to Metabolic Health. Front Endocrinol (Lausanne). 2022 Jun 29;13:892677. doi: 10.3389/fendo.2022.892677. eCollection 2022. PMID 35872982
- [Derived] Fritsche A, Wagner R, Heni M, Kantartzis K, Machann J, Schick F, Lehmann R, Peter A, Dannecker C, Fritsche L, Valenta V, Schick R, Nawroth PP, Kopf S, Pfeiffer AFH, Kabisch S, Dambeck U, Stumvoll M, Bluher M, Birkenfeld AL, Schwarz P, Hauner H, Clavel J, Seissler J, Lechner A, Mussig K, Weber K, Laxy M, Bornstein S, Schurmann A, Roden M, de Angelis MH, Stefan N, Haring HU. Different Effects of Lifestyle Intervention in High- and Low-Risk Prediabetes: Results of the Randomized Controlled Prediabetes Lifestyle Intervention Study (PLIS). Diabetes. 2021 Dec;70(12):2785-2795. doi: 10.2337/db21-0526. Epub 2021 Sep 16. PMID 34531293
- See also: Click here for more information about this study: research in the DZD --> klinische Studien — http://www.dzd-ev.de